CLINICAL TRIAL: NCT01239667
Title: Rehabilitative Care to Patients With Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College Absalon (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Johny Lauritsen, University College Sjaelland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: pla123
Record Dates: First submitted 2010-10-25; First posted 2010-11-11 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2010-10

CONDITIONS: Rehabilitation After Heart Failure
Keywords: Health related quality of Life, Self Care behavior, activities of daily living

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Life style counseling (Experimental): Individual oriented rehabilitation plan in collaboration with the patient followed by measuring health related quality of life and self care behavior
  Interventions: Other: Individual oriented planning of the rehabilitation program for patients with heart failure

INTERVENTIONS:
Other: Individual oriented planning of the rehabilitation program for patients with heart failure — Individual oriented rehabilitation plan in collaboration with the patient followed by measuring health related quality of life and self care behavior

SUMMARY:
Hypothesis and objectives of the study Systematic preparation of rehabilitation plan for rehabilitation in Phase III based on identification of self-care behavior patients with heart failure in NYHA class II and III, leading to patients' self-care behaviors strengthened, which will result in increased health status and ADL level 6 months after discharge from hospital with heart failure .

Target

1. To develop evidence-based clinical guidelines for patient rehabilitation phase III
2. To test the effect of individual rehabilitation plans based on clinical guidelines for patient rehabilitation in Phase III. Efficacy evaluated in relation to changes in self-care behaviors, health status and ADL function.

Material and Methods:

Controlled longitudinal study. Each intervention patient receives before the end of hospital rehabilitation designed a specific rehabilitation plan also contacted the patient by specially trained nurse telephone 4 and 12 weeks after completion of their rehabilitation in hospital and the patient has the opportunity to contact the department when needed. The effect of rehabilitation assessed by sending questionnaires SF 36 and EHFScB Scale 9, to assess patients' ADL functioning, self-care behaviors and self-rated health.

All patients participating in the planned rehabilitation in hospitals, so that the baseline is the end of Phase II. Intervention based on an analysis of the individual's need for continued rehabilitation (self care behavior, health status, ADL function) and the patient's perception of own situation. Draw up a plan and program together with the patient

DETAILED DESCRIPTION:
Rehabilitation for people with serious illness, has been in focus over the last 10-15 years which is also valid for heart field (1). The focus of cardiac rehabilitation has been on the efficacy of treatment in relation to mortality, morbidity and health-related quality of life (HRQoL).

Purpose of rehabilitation are:

"Rehabilitation is a targeted and time-bound collaborative process between an individual, relatives and professionals. The aim is that citizens who have or are at risk of significant limitations in physical, mental and / or social functioning, achieve an independent and meaningful life. Rehabilitation based on the citizen's whole life situation and decisions made by a coordinated, coherent, knowledge-based action (1).

Background. Worldwide, estimated that around. 50 million people suffer from heart disease (2). In Denmark assumed that 60,000 people live with chronic heart failure, with prevalence increasing with increasing age (3) (4). In 2005 there were 142,245 hospitalizations with cardiovascular disease in Denmark, by 86,336 people, 1,786 per 100,000 men and 1,409 per 100,000 women. Viewed in isolation on heart-related deaths in the period 1998 -2005 is a decrease in mortality in general, and in 30 day mortality after AMI decreased from 10 to 4% (5). Cardiac rehabilitation has been made in traditional hospital setting and there is a documented effect of effort in terms of patients' physical function, decrease in relapse of disease, and decrease in morbidity and mortality (2) (6) (7) (8) (9).

Hypothesis and objectives of the study Hypothesis: Systematic preparation of rehabilitation plan in Phase III based on the identification of self care behavior patients with heart failure in NYHA class II and III, leading to patients' self-care behaviors strengthened, which will result in improved health status and ADL level 6 months after discharge from hospital with heart failure .

Target

1. To develop evidence-based protocol for patient rehabilitation phase III
2. To test the effect of individual rehabilitation plans based on evidence-based knowledge of patient rehabilitation in Phase III. Efficacy evaluated in relation to changes in self-care behaviors, health status and ADL function.

Materials and methods. 3.1 Population: Patients recruited from Zealand Region Hospital South in Naestved and Slagelse. There are printed annually 55-60 patients with heart failure from each of the respective hospitals. The material in the study are women and men with heart failure in NYHA class II - III of participants are calculated based on strength calculation.

Inclusion:

Patients in NYHA II-III Participation happens after written informed consent. Patients included in the respective intervention or control group depending on the hospital site.

Exclusion:

Patients who do not wish to participate. Patients with language and communication impedes Sufficient participation. Patients who do not understand information, as well as patients diagnosed with neurological deficits.

Calculation of sample size:

Calculation of patient numbers are based on strength calculation. The level of type 1 error set at 5% and type 2 errors to 20%, and expected an improvement in ADL level at 50%, Power Calculation shows that the participating 60 patients in the control and 60 patients in the intervention group (http:/ / statpages.org / proppowr.html). With an expected dropout rate of 25%, therefore, invited 72 patients in each group

Design. quasi experimental study of patients from the Regions Hospital in Naestved and the hospital in Slagelse. Each intervention patient receives before the end of hospital rehabilitation designed a specific rehabilitation plan also contacted the patient by specially trained nurse telephone 4 and 12 weeks after completion of their rehabilitation in hospital and the patient has the opportunity to contact the department when needed. The effect of rehabilitation assessed by sending questionnaires SF 36 and EHFScB Scale 9 (36) to assess patients' ADL functioning, self-care behaviors and self-rated health. Patients included in the experimental and control group. Randomization and blinding is not possible since the staffing resources are not sufficient to enable the staff only have contact with the respective intervention or control patients.

All patients participating in the planned rehabilitation in hospitals, so that the baseline is the end of Phase II. Intervention based on an analysis of the individual's need for continued rehabilitation (selfcare behavior, health status, ADL function) and the patient's perception of own situation. Draw up a plan and program together with the patient. The program must be tailored to the individual patient's possibilities. The program supplied with guides to what the patient can do yourself. The patient acknowledged copy of the plan to your physician and home care. Furthermore, the patient will be contacted by specially trained nurse telephone 4 and 12 weeks after initiation of phase III rehabilitation, providing telephone support from a structured interview guide. Patients also have the opportunity outside the agreed times to contact the specialist nurse.

Variables: Demographic data, sex, age, living alone, dependent / independent of help from others, diagnosis, status of job, comorbidities, NYHA class

NYHA classification is carried out by specialists at discharge from hospital and transition to rehabilitation

Self-Care Behavior and ADL functions, estimated using the European Heart Failure Self-Care Behavior Scale. The instrument is translated and face validated in a pilot test before use. The test measures patients' ability to assess their own situation and ability to act on the observations made (36).

Health Status Assessed with Short Form 36 (SF-36). The form is generic and covers the patient's perception of their health. SF-36 has been translated into Danish and validated (37). SF-36 includes 36 questions on self-assessment of health status that includes eight specific areas: physical functioning, physical constraints, pain, general health, energy / fatigue, social functioning, psychological constraints and psychological wellbeing. For each of the eight strands transformed responses to an interval scale from 0-100 where 0 indicates no impairment or full restriction and 100 indicates full function or no restriction.

Process variable: compliance over nursing program examined self-reported data.

Statistical analysis:

Data will be analyzed in the statistical program SPSS. Ratio-scaled data from the two groups is tested by F test MHP. of distribution. For normally distributed data are compared by using parametric methods (t test), otherwise non-parametric methods (Mann-Whitney Rank Sum Test). Nominal Scale Data compared by chi-square test or by using 95% confidence interval.

The project reported to the Data Inspectorate. Furthermore, the experiment reported to the local Research Ethics Committee, and to www.Clinicaltrials.gov so that rights to the project ensured.

.

ELIGIBILITY:
Inclusion Criteria:Patients who are 18 years or older and valued at NYHA II and III are included in the study. -

Exclusion Criteria:

* Patients who do not wish to participate. Patients with language and communication impedes Sufficient participation. Patients who do not understand information, as well as patients diagnosed with neurological deficits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-05 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Health related quality of life | Measured 6 month after discharge from hospital
  Evidence for health related quality of life in heart failure patients in the rehabilitation phase, measured with instrument SF 36
Self Care Behavior | measured 6 month after discharge
  Mesure the patients self care behavior by using the instrument European Heart Failure Self Care Behavior Scale
Activities of Daily Living | 6 month after discharge
  measure the patients PADL and IADL functions

CONTACTS AND LOCATIONS:
Overall Officials: Palle Larsen, MSN and Ph.d. student, Principal Investigator — Univcersity College Sjaelland
Locations (1):
- University of Aarhus Denmark, Aarhus, Aarhus, Denmark